CLINICAL TRIAL: NCT00049699
Title: A Phase I Trial of VNP40101M, a Novel Alkylating Agent, Administered Weekly for Patients With Advanced or Metastatic Cancer
Brief Title: VNP40101M in Treating Patients With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: VION-CLI-028; CDR0000258355 (Registry Identifier: PDQ (Physician Data Query)); YALE-HIC-16775
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2004-03

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; small intestine lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; unspecified adult solid tumor, protocol specific; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — laromustine

INTERVENTIONS:
Drug: laromustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of VNP40101M in treating patients who have advanced or metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxic effects of VNP40101M in patients with advanced or metastatic solid tumor or lymphoma.
* Determine the maximum tolerated dose of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the antitumor effects of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive VNP40101M IV over 15 minutes on days 1, 8, and 15. Treatment repeats every 28 days.

Cohorts of 3-6 patients receive escalating doses of VNP40101M until the maximum tolerated dose is determined.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced or metastatic solid tumor or lymphoma for which no curative or standard effective therapy exists
* Measurable or evaluable disease
* Primary brain tumors or brain metastases allowed provided neurologic deficits are stable and do not preclude study compliance

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 3 months

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hematocrit at least 30% (transfusion allowed)
* No bleeding diathesis

Hepatic

* PT and PTT no greater than 1.5 times the upper limit of normal (ULN)
* Bilirubin no greater than 1.5 times ULN
* ALT and AST no greater than 1.5 times ULN (3 times ULN if liver metastases present)
* Albumin at least 2.5 gm/dL

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* At least 3 months since prior myocardial infarction
* No symptomatic coronary artery disease
* No arrhythmias requiring medication
* No uncontrolled congestive heart failure

Pulmonary

* No dyspnea on minimal or moderate exertion
* DLCO and FEV1 at least 60% predicted

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled active bleeding (e.g., active peptic ulcer disease)
* No active infection
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Recovered from acute toxicities of prior biologic therapy (persisting, chronic toxicity allowed if stable and no greater than grade 1)

Chemotherapy

* More than 6 months since prior high-dose chemotherapy with stem cell support
* More than 3 weeks since prior cytotoxic chemotherapy (6 weeks for mitomycin or nitrosoureas)
* Recovered from acute toxicities of prior chemotherapy (persisting, chronic toxicity allowed if stable and no greater than grade 1)

Endocrine therapy

* At least 2 weeks since prior hormonal therapy

Radiotherapy

* Recovered from acute toxicities of prior radiotherapy (persisting, chronic toxicity allowed if stable and no greater than grade 1)

Surgery

* At least 2 weeks since prior surgery

Other

* No other concurrent standard or investigational treatment for cancer
* No concurrent disulfiram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (3):
- United States (3):
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Veterans Affairs Medical Center - West Haven, West Haven, Connecticut
  - Ireland Cancer Center, Cleveland, Ohio